CLINICAL TRIAL: NCT02934399
Title: Dynamic Hormone Diagnostics (Ultradian)
Brief Title: Dynamic Hormone Diagnostics in Endocrine Disease
Acronym: ultradian
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Karolinska Institutet (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Evaggelismos Hospital, Greece (Unknown)
Responsible Party: Sponsor
Other Study IDs: REKno 2015/872
Record Dates: First submitted 2016-01-12; First posted 2016-10-17 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2020-08

CONDITIONS: Adrenal Insufficiency; Congenital Adrenal Hyperplasia; Cushing Syndrome; Growth Hormone Deficiency; Acromegaly; Primary Hyperaldosteronism
Keywords: dynamic hormone diagnostics; adrenal insufficiency; congenital adrenal hyperplasia; primary hyperaldosteronism; cushing syndrome; growth hormone deficiency; acromegaly
MeSH Terms: conditions — Adrenal Insufficiency; Adrenal Hyperplasia, Congenital; Cushing Syndrome; Dwarfism, Pituitary; Acromegaly; Hyperaldosteronism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Subcutaneous fluid/dialysate, saliva samples, urine samples and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Healthy controls (HC): Definition of the normal circadian and ultradian profiles of pituitary and adrenal hormones in healthy subjects:Each subject (total number 200, anticipated 50 per study centre) will be sampled by the ULTRADIAN sampling device for 27 hours. Day to day hormonal variability:A subgroup of 20 subjects will be asked to undergo sampling on three occasions to assess reproducibility of hormonal levels over time. Comparison of tissue and blood concentrations of hormones: 20 subjects will be asked to participate in the study comparing hormonal tissue level and blood levels.
  Interventions: Other: 27 hour subcutaneous fluid sampling
- Cushing syndrome (CS): Diagnosis of Cushing's syndrome by ULTRADIAN dynamic cortisol measurements The primary objective is to establish circadian and ultradian hormonal profiles of patients with Cushing's from 24 hour ambulatory sampling of subcutaneous fluid.
  A secondary aim is to compare the pre and post-operative hormonal profiles of patients with Cushings and to compare these results to age/sex matched control
  Study subjects: Subjects with established clinical and biochemical Cushing's syndrome (ACTH-producing pituitary adenoma or ACTH-independent adrenal source).
  Interventions: Other: 27 hour subcutaneous fluid sampling
- Adrenal insufficiency (AI): Monitoring of adrenal insufficiency (AI) by ULTRADIAN dynamic cortisol and ACTH measurements Aims and objectives: to compare hormonal profiles of patients with Adrenal insufficiency on conventional replacement regimes to age/sex matched controls.
  Study subjects: Subjects with established primary (adrenal) AI
  Interventions: Other: 27 hour subcutaneous fluid sampling
- Congenital adrenal hyperplasia (CAH): Monitoring of congenital adrenal hyperplasia (CAH) by ULTRADIAN dynamic cortisol, ACTH, and androgen measurements Aims and objectives: to compare hormonal profiles of patients with CAH on conventional replacement regimes to age/sex matched controls.
  Study subjects: Individuals with established CAH either salt- wasting or simple virilisation forms on glucocorticoid replacement therapy
  Interventions: Other: 27 hour subcutaneous fluid sampling
- Primary hyperaldosteronism (PHA): Diagnosis of primary hyperaldosteronism (PHA) by ULTRADIAN dynamic aldosterone and renin measurements Aims and objectives: The primary objective is to establish circadian and ultradian profiling of free aldosterone and renin in subcutaneous tissue.
  Secondary objectives are (1) to compare pre and post-operative profiles (2) to identify profiles typical for adenoma as opposed to bilateral hyperplasia and (3) to compare profiles to age/sex matched controls.
  Study subjects: Subjects with suspected PHA.
  Interventions: Other: 27 hour subcutaneous fluid sampling
- Growth hormone insufficiency (GHD): Diagnosis of growth hormone deficiency (GHD) by ULTRADIAN dynamic growth hormone measurements Aims and objectives: The primary objective is to establish hormonal circadian and ultradian profiles of adult GHD by analysing the growth hormone profile in the subcutaneous tissue fluid.
  Study subjects: Adult subjects with established clinical and biochemical GHD.
  Interventions: Other: 27 hour subcutaneous fluid sampling
- Acromegaly (A): Diagnosis and treatment of acromegaly by ULTRADIAN dynamic growth hormone measurements Aims and objectives: The primary objective is to establish hormonal profiles of patients with Acromegaly A secondary objective is to compare pre and post-operative profiles and to compare these profiles to age/sex matched controls.
  Study subjects: Patients with established clinical and biochemical Acromegaly by current diagnostic criteria
  Interventions: Other: 27 hour subcutaneous fluid sampling

INTERVENTIONS:
Other: 27 hour subcutaneous fluid sampling — One hour prior to the microdialysis catheter insertion the participants will be asked to receive a local anaesthetic on the injection site for the microdialysis catheter. Lignocaine 1% will be injected subcutaneously at a localised site on the abdomen covering a horizontal area of about 5cm after a brief acclimatisation period at the hospital.
  A sterile linear catheter will be inserted using aseptic precautions at the anaesthetised site on the abdomen. The catheter is connected at one end to the microdialysis pump, and at the other end to the automated collection device. Subcutaneous tissue microdialysis samples will be collected regularly for the duration of the sampling period (27 hours).

SUMMARY:
The study will investigate 27 hour profiles of hormones in the subcutaneous tissue of healthy subjects and patients with Addison's, Congenital Adrenal Hyperplasia, Growth Hormone Deficiency, acromegaly, Cushings and Primary Hyperaldosteronism during conventional diagnostic and therapeutic follow-up.

The 27 hour monitoring by ULTRADIAN takes into account the rhythm of hormones throughout the day. It is hoped that this information may in the future improve and simplify diagnostic procedures. Follow-up of patients in endocrinology still remains difficult including clinical signs of over and under-treatment, questionnaires of quality of life and blood testing necessitating often retesting. Simplification of the diagnostic procedure by obtaining detailed knowledge about the rhythm of hormones may contribute to the improvement and individualization of treatment and may decrease morbidity and mortality of endocrine patients.

DETAILED DESCRIPTION:
Microdialysis fluid will be collected from all participants using the ULTRADIAN dynamic diagnostics system. This is a 3-component collection system which can easily be attached to a belt and allows participants to continue with their normal everyday activities whilst undergoing sampling. The micro-fractions are minute, the volume would normally be by far too small to use with current immunoassays.

ULTRADIAN will overcome this hurdle by introducing two novel techniques; ultrasensitive liquid chromatography tandem mass spectroscopy (LCMS/MS) for steroid hormones, and the proximity extension assay (PEA®), which allows the simultaneous assay of up to 96 analytes in only 1 µL fluid.

The microdialysis sampling will be performed in addition to the conventional diagnostic sampling, and during normal follow-up of patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18-68 years, non-smokers or regular smokers of greater than 6 cigarettes a day, BMI 16-29
* Male and female Cushing's syndrome aged 18-68 years with biochemically confirmed based on cortisol and ACTH measurements, dexamethasone suppression test and 1 of the following positive investigations (24 hour urine cortisol, salivary/serum cortisol profile). Visible tumour in the pituitary and/or one of the following positive tests pointing to pituitary source for ACTH overproduction (bilateral petrosal sinus sampling, corticotropin releasing hormone test, high dose dexamethasone suppression test) or adrenal tumour considered fit for surgery. No contraceptives for 6 weeks prior to sampling (females only). Patients on medical therapy e.g. metyrapone for Cushings to have a 2 week washout off treatment prior to sampling
* Male and female aged 18 -68 years with biochemically confirmed adrenal insufficiency based on basal cortisol and ACTH measurements and/or Synacthen test +/- adrenal antibodies, and on oral hydrocortisone or cortisone acetate glucocorticoid replacement therapy
* Female aged 18-68 years with biochemically confirmed salt-wasting or simple virilising CAH based on 17OHP, cortisol, androgen, renin and ACTH measurements; disease causing mutation in CYP21A2 and/or synacthen testing.
* Male and female subjects aged 18 -68 years with biochemical confirmation of PHA based on a valid pathological aldosterone/renin ratio and non-suppressible aldosterone levels on one of the currently used confirmatory tests (saline/oral fludrocortisone test). Unilateral only - diagnostic CT and/or adrenal vein sampling
* Male and female subjects aged 18-68 years with biochemically confirmed GHD (arginine growth hormone releasing hormone test, insulin tolerance test, known pituitary disease with confirmed pan hypopituitarism)
* Male and female aged 18-68 years with biochemically confirmed acromegaly (oral glucose tolerance test or GH day curve and diagnostic insulin growth factor 1 levels) with radiological evidence of a pituitary adenoma.

Exclusion Criteria:

* Healthy controls undergoing or planning pregnancy or lactating women. Presence of any unstable pathological condition in past 3 months. On any regular prescribed medications (except contraception). Prior or current history of an endocrine disorder. Known allergy to Lignocaine, plasters. Current or past steroid therapies (oral, inhaled, parenteral or topical) or other interfering medication in last 3 months. Regular alcohol intake great then 26units of alcohol per week.Taking of any investigational drug within the past two months. Abuse of illicit drugs. Occasional smokers of cigarettes not able to abstain for sampling period or smoking less than 6 cigarettes a day. Needle phobia. Interfering diet/over the counter herbal remedies in last 14 days.
* Cushing syndrome: Undergoing or planning pregnancy (females only). Known allergy to Lignocaine. Adrenal cancer (post-operative histology diagnosis),cyclic Cushings, squamous cell lung carcinoma, bronchial carcinoid and occult ectopic Cushings. Concurrent use of steroid therapy for any other medical condition (oral, inhaled, parenteral or topical)
* Adrenal insufficiency: Undergoing or planning pregnancy, known allergy to Lignocaine, use of other steroid medications other than their standard glucocorticoid and fludrocortisone replacement, other interfering medication or diet within 2 weeks of sampling.
* CAH: Males, females undergoing or planning pregnancy, known allergy to Lignocaine, use of other steroid medications other than their standard glucocorticoid and fludrocortisone replacement or other interfering medication or diet within 2 weeks of sampling
* Primary hyperaldosteronism: Undergoing or planning pregnancy (females only), known allergy to Lidocaine, known adrenal failure and/or on steroid therapy (oral, inhaled, parenteral or topical), concurrent use of interfering medication ( i.e. specific interfering antihypertensive medication) or diet within 2-4 weeks of ultradian sampling
* GHD: Undergoing or planning pregnancy (females only) or known allergy to Lignocaine
* Acromegaly: Undergoing or planning pregnancy (females only), known allergy to Lignocaine treatment with somatostatin analogues and other interfering medication (e.g. oestrogens)

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Controls and patients with established Cushing syndrome, Adrenal Insufficiency, Congenital adrenal hyperplasia, Primary hyperaldosteronism, Acromegaly and Growth hormone deficiency
Sampling Method: Probability Sample
Enrollment: 528 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
steroids | 27 hours
  Physiological hormonal curve by sampling of 27h subcutaneous fluid to measure steroids
androgens | 27 hours
  Physiological hormonal by sampling of 27h subcutaneous fluid to measure androgens
mineralocorticoids | 27 hours
  Physiological hormonal curve by sampling of 27h subcutaneous fluid to measure mineralocorticoids
ACTH | 27 hours
  Physiological hormonal curve by sampling of 27h subcutaneous fluid to measure ACTH
growth hormone | 27 hours
  Physiological hormonal curve by sampling of 27h subcutaneous fluid to measure growth hormone
steroids in Addison disease | 27 hours
  Hormonal curve by sampling of 27h subcutaneous fluid to measure steroids
steroids in congenital adrenal hyperplasia | 27 hours
  Hormonal curve by sampling of 27h subcutaneous fluid to measure steroids
androgen in congenital adrenal hyperplasia | 27 hours
  Hormonal curve by sampling of 27h subcutaneous fluid to measure androgens
growth hormone in acromegaly | 27 hours
  Hormonal curve by sampling of 27h subcutaneous fluid to measure growth hormone
growth hormone in growth hormone deficiency | 27 hours
  Hormonal curve by sampling of 27h subcutaneous fluid to measure growth hormone
mineralocorticoids in primary hyperaldosteronism | 27 hours
  Hormonal curve by sampling of 27h subcutaneous fluid to measure mineralocorticoids

SECONDARY OUTCOMES:
Intra-individual variability and the accuracy of steroids hormones | 27 hours
  comparison of steroids levels in repetitive testing
Intra-individual variability and the accuracy of androgens | 27 hours
  comparison of androgens levels in repetitive testing
Intra-individual variability and the accuracy of mineralocorticoids | 27 hours
  comparison of mineralocorticoids levels in retesting by microdialysis
Intra-individual variability and the accuracy of growth hormone | 27 hours
  comparison of growth hormone levels in retesting by microdialysis
Intra-individual variability and the accuracy of ACTH | 27 hours
  comparison of ACTH levels in retesting by microdialysis

CONTACTS AND LOCATIONS:
Overall Officials: Stafford Lightman, Professor, Principal Investigator — University of Bristol; Sophie Bensing, MD phD, Principal Investigator — Karolinska Institutet; Stylianos Tsagarakis, Professor, Principal Investigator — Evaggelismos Hospital
Locations (4):
- Evangelissmos hospital, Athens, Greece
- Haukeland University Hospital, Bergen, Norway
- Karolinska Institutet, Stockholm, Sweden
- Bristol University hospital, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Upton TJ, Zavala E, Methlie P, Kampe O, Tsagarakis S, Oksnes M, Bensing S, Vassiliadi DA, Grytaas MA, Botusan IR, Ueland G, Berinder K, Simunkova K, Balomenaki M, Margaritopoulos D, Henne N, Crossley R, Russell G, Husebye ES, Lightman SL. High-resolution daily profiles of tissue adrenal steroids by portable automated collection. Sci Transl Med. 2023 Jun 21;15(701):eadg8464. doi: 10.1126/scitranslmed.adg8464. Epub 2023 Jun 21. PMID 37343084